CLINICAL TRIAL: NCT00177463
Title: A Pilot Add-on Randomized, Placebo Controlled Intervention Trial of Cognitive Enhancement in Persons With Bipolar Disorder Using an Antioxidant and Advanced Glycation End (AGE) Product Inhibitor: L-Carnosine
Brief Title: L-Carnosine for Bipolar I Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, K.N. Roy Chengappa, Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Chengappa L-carnosine; IRB #0410144
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Bipolar I Disorder
Keywords: L-carnosine; Bipolar I disorder; Cognitive enhancement
MeSH Terms: interventions — Carnosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L- Carnosine (Experimental): an antioxidant and AGE inhibitor, 500 mg/day, increasing each week in titration reaching 2000 mg/day in 4 weeks and maintained for rest of trial
  Interventions: Drug: L-carnosine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: L-carnosine

INTERVENTIONS:
Drug: L-carnosine — an antioxidant and AGE inhibitor, 500 mg/day, increasing each week in titration reaching 2000 mg/day in 4 weeks and maintained for rest of trial
  Other Names: L Carnosine

SUMMARY:
Our hypothesis is that oral L-carnosine treatment (as compared with placebo) will enhance cognitive abilities (specifically: measures of attention, executive function, working memory, visuospatial ability and language) in persons with bipolar disorder. Secondarily, we hypothesize there will be secondary improvements in positive, negative and mood symptoms with L-carnosine treatment.

We aim to test these hypotheses by conducting a randomized, placebo controlled, add on treatment trial of L-carnosine (added to existing antipsychotic treatment) on 48 recruited subjects with DSM IV TR bipolar disorder for a period of 12 weeks. Measures of cognition, and psychopathology will be utilized for evaluating primary and secondary outcomes, along with safety assessments.

DETAILED DESCRIPTION:
OBJECTIVE:

It is our hypothesis that L-carnosine treatment of persons with bipolar illness will improve their cognitive outcomes, more specifically, measures of attention and executive function, verbal and visuospatial memory and psychomotor performance, relative to placebo treatment. We also hypothesize that L-carnosine treatment may secondarily improve any residual affective symptoms.

RESEARCH PLAN:

We aim to test these hypotheses by conducting a randomized, placebo controlled, add on treatment trial of L-carnosine (added to ongoing prescribed pharmacological treatment, for example - lithium, anticonvulsants, antipsychotic agents and depressants) for a period of 12 weeks. Measures of cognition, and psychopathology will be utilized for evaluating primary and secondary outcomes, along with safety assessments.

METHODS:

Up to 48 subjects with DSM IV TR bipolar I disorder will be recruited from Western Psychiatric Institute and Clinic, Mayview State Hospital and Mon Yough Community Services, Inc. using a 1:1 randomization, subjects who sign a informed consent document will be randomized to receive L-carnosine or placebo.

It is expected that 12 of the 48 subjects may not meet inclusion/exclusion criteria, leaving 36 consenting adults (18 to 65 years) with DSM IV-TR Bipolar Disorder who will be assessed for euthymia (Young Mania Rating Scale Score ≤ 10, Montgomery Asberg Depression Rating Scale Score of ≤ 10) over a one month period (2 assessments) while receiving stable doses of their current medications. They will also be assessed for cognitive dysfunction (attention/executive function, immediate and declarative memory, and psychomotor performance) using Cogtest - a proprietary neuropsychological library of 19 tests. These subjects will be characterized for normal pre-morbid IQ, no ECT treatment in past 6 months, no alcohol or substance dependence in past 6 months, mini-mental state score ≥ 24.

L-carnosine (or placebo) will be administered using random assignment at a dose of 500 mg/day, increasing each week by 500 mg to a dose of 2000 mg/day (twice daily schedule) in 4 weeks; as an adjunct to existing psychotropic medicines. The dose of 2000 mg (or less, i.e. a minimum of 500 mg if tolerability is an issue) will be continued for 8 additional weeks. L-carnosine is not known to have interactions with psychotropic drugs but mood-stabilizer levels will be monitored.

Standard psychopathology rating scales will be administered to evaluate secondary aims such as impact on residual symptoms of bipolar disorder. Safety will be assessed by tailing a careful medical history and physical examination at screening and evaluating results of laboratory measures. Any adverse effects will be assessed by asking questions at each visit, and if required bring subjects in for assessments outside the scheduled visits, and by telephone contact in between longer scheduled visits.

SIGNIFICANCE:

Cognitive dysfunction can seriously hinder improved functional outcomes in persons with schizophrenia or bipolar disorder. If this short term intervention with L-carnosine shows promise, more definitive studies using adequate powered sample sizes, and of longer duration can be conducted. If improvements in cognitive problems are linked to improved functional outcomes using such supplemental treatments, an important therapeutic milestone in bipolar disorder will have been achieved.

ELIGIBILITY:
Inclusion Criteria:

* DSM IV - TR diagnosis of bipolar I disorder or
* Ages 18 to 65 years
* Men or Women
* Ability to read and communicate in English
* 8th grade education or greater
* Ability to provide informed, competent and written consent
* Current medication and mood status (Y-MRS and MADRS scores less than or equal to 10) is stable for greater than or equal to 4 weeks.

Exclusion Criteria:

* Medically unstable conditions
* Known allergy to L-carnosine
* Current cognitive decline is attributable to a diagnosis of dementia or other neurological disorder, including HIV dementia or cognitive decline
* Pregnant or lactating women
* Mini-mental state examination score (MMSE) less than or equal to 23.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
That L-carnosine treatment of persons with bipolar illness will improve their cognitive outcomes, specifically, measures of attention and executive function, verbal and visuospatial memory and psychomotor performance, relative to placebo treatment. | 12 weeks treatment

SECONDARY OUTCOMES:
That L-carnosine treatment may secondarily improve any residual affective symptoms in subjects with bipolar disorder. | 12 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: K.N. Roy Chengappa, MD, Principal Investigator — Western Psychiatric Institute and Clinic
Locations (3):
- United States (3):
  - Mayview State Hospital, Bridgeville, Pennsylvania
  - Mon-Yough Community Services, Inc., McKeesport, Pennsylvania
  - Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Connect to NARSAD list of active research studies — http://www.narsad.org/